CLINICAL TRIAL: NCT06331312
Title: A Multi-center, Open-label Extension Study of Subcutaneous Secukinumab to Evaluate the Long-term Safety and Tolerability in Polymyalgia Rheumatica (PMR)
Brief Title: Open-label, Long-term Safety Study of Secukinumab in Polymyalgia Rheumatica (PMR)
Acronym: REPLENISH-EXT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457C22301E1; 2023-508077-85-00 (Other: EU CT number)
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Polymyalgia Rheumatica
Keywords: Polymyalgia Rheumatica (PMR); secukinumab; monoclonal antibody; subcutaneous (s.c.); extension; long-term; safety; REPLENISH
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Secukinumab 300mg (Experimental): All eligible participants will receive secukinumab 300 mg s.c. (2 x 150mg/1mL PFS secukinumab) from baseline and every 4 weeks up to 2 years. The study medication may be modified/adjusted after the initial doses of 300mg s.c. (decreased to 150mg s.c. q4w or increased again from 150mg s.c. q4w to 300mg s.c. q4w) if deemed appropriate by the investigator. Dose modification/adjustment may only occur from Week 24 visit onwards. The modification/adjustment of the study medication will be determined at a site visit.
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: Secukinumab — 2 x 150mg/1mL PFS secukinumab

SUMMARY:
The purpose of this extension study is to assess the safety and tolerability of secukinumab when administered long-term in patients with polymyalgia rheumatica.

DETAILED DESCRIPTION:
The study will consist of an up to 4-week screening period, an up to 2-year Treatment Period which includes two Treatment Periods, and a 16-week treatment-free follow-up period (20 weeks post last dose of secukinumab).

Treatment period:

There will be two Treatment Periods (TPs): TP1 will be from the first dose administration of secukinumab (Baseline) to Week 24, where visits will occur every 4 weeks, and TP2 will be from post Week 24 visit (post-dose) to up to 2 years. Participants will return to the study site every 4 weeks from Baseline until Week 24 (Weeks 16 and 20 visits are optional on-site visits and needed when participants are unwilling/uncomfortable to self-administer study treatment at home/offsite), then every 12 weeks afterwards in TP2 for resupply of study medication but may return earlier if needed (i.e., those participants who are unwilling/uncomfortable to self-administer study treatment can continue to visit site every 4 weeks for drug administration if they wish to do so).

Follow-up period: An EoS visit (20 weeks after last administration of secukinumab) will be done for all participants, regardless of whether they complete the entire study as planned, or they discontinue prematurely.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed 52-week Treatment Period as per protocol in a Novartis study of secukinumab in PMR patients (the "core study" - Study CAIN457C22301), AND

  * who have experienced a relapse during the treatment-free follow-up period of the core study, AND
  * who have not been on rescue treatment.
* The participant would potentially derive benefit from secukinumab, and the benefit outweighs the risk, based on the investigator's judgement.

Exclusion Criteria:

* Use of prohibited medications, as specified in the protocol
* History of ongoing, chronic or recurrent infectious disease (i.e., human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV), active tuberculosis infection (TB))
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for basal cell carcinoma or actinic keratosis that have been treated with no evidence of recurrence in the past 3 months carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
* Live vaccinations (e.g., monkey pox vaccine, oral polio vaccine, varicella/zoster vaccines) within 6 weeks prior to Baseline
* Subjects whose participation in the extension study could expose them to an undue safety risk

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2028-08-22 (Estimated); Study Completion 2028-08-23 (Estimated)

PRIMARY OUTCOMES:
Incidences of treatment emergent adverse events (AEs) and serious adverse events (SAEs) | After the first dose of study treatment and within 84 days after the last dose
  The number and percentage of participants with treatment emergent AEs/SAEs will be summarized. No hypothesis testing will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (107):
- United States (19):
  - Arizona Arthritis and Rheumatology Associates PLLC, Avondale, Arizona
  - Sun Valley Arthritis Center Ltd, Peoria, Arizona
  - Orrin Troum MD and Medical Associates, Santa Monica, California
  - Center for Rheumatology Research, West Hills, California
  - Millennium Clinical Trials, Westlake Village, California
  - Rheumatology Associates of South Florida, Boca Raton, Florida
  - UF Health Cancer Center, Gainesville, Florida
  - Sarasota Arthritis Res Ctr, Sarasota, Florida
  - West Broward Rheumatology Associates Inc, Tamarac, Florida
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - Klein and Associates, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Clinical Research Inst of MI, Saint Clair Shores, Michigan
  - Kansas City Physician Partners, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Paramount Med Rsrch and Consult LLC, Middleburg Heights, Ohio
  - Prolato Clinical Research Center, Houston, Texas
  - Accurate Clinical Research Inc, San Antonio, Texas
  - Advanced Rheumatology of Houston, Spring, Texas
- Argentina (2):
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (3):
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Heidelberg Heights, Victoria
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Brazil (3):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Novartis Investigative Site, Québec, Quebec, Canada
- Chile (2):
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
- Colombia (3):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Cali, Valle del Cauca Department
- Czechia (6):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hlučín
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
  - Novartis Investigative Site, Zlín
- Denmark (3):
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Gandrup
  - Novartis Investigative Site, Vejle
- France (12):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Cholet
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (7):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Rendsburg
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Ramat Gan, Israel
- Italy (5):
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Emilia, RE
- Japan (14):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Ōme, Tokyo
  - Novartis Investigative Site, Shimonoseki, Yamaguchi
  - Novartis Investigative Site, Chūō, Yamanashi
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Beirut, Lebanon
- Novartis Investigative Site, Guadalajara, Jalisco, Mexico
- Netherlands (3):
  - Novartis Investigative Site, Almelo, Overijssel
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Groningen
- Poland (3):
  - Novartis Investigative Site, Bytom
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Cape Town, Western Cape, South Africa
- Spain (7):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Sankt Gallen
- United Kingdom (3):
  - Novartis Investigative Site, Barnet
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com